CLINICAL TRIAL: NCT06657001
Title: Enabling Microbiomics- Driven Personalized Nutrition (EMPOWER)
Brief Title: Enabling Microbiomics- Driven Personalized Nutrition
Acronym: EMPOWER
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, Principal Investigator, Mayo Clinic
Other Study IDs: 24-007049
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Disease (IBD); Irritable Bowel Syndrome (IBS); Celiac Disease; Diarrhea; Constipation; Microbiome; Crohn's Disease; UC - Ulcerative Colitis; Microscopic Colitis; Functional Dyspepsia
Keywords: GI Disorders; Microbiomics; Diet; Microbiome; Nutrition; GI Function
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Celiac Disease; Diarrhea; Constipation; Crohn Disease; Colitis, Ulcerative; Colitis, Microscopic; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GI Disorders: Inflammatory Bowel Disease, Irritable Bowel Syndrome, Crohn's Disease, Celiac Disease, Diarrhea, Constipation

SUMMARY:
The goal of this observational research study is to determine how diet contributes to various gastrointestinal related conditions.

The main question investigators aim to answer is:

Are host genetics, diet, and microbiome all important determinants of GI disorders, and how their relative contribution varies among individuals and populations.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Gastrointestinal patients with or without genomic sequencing results available for the following cohorts:

  * Inflammatory Bowel Disease (IBD)
  * Irritable Bowel Syndrome (IBS)
  * Crohn's Disease
  * Celiac Disease
  * Diarrhea
  * Constipation
* Healthy age and sex matched controls with or without genomic sequencing results available

  o Control is defined as patients without gastrointestinal disease or no symptoms at time of sampling
* Able to provide written, informed consent
* Participant has a smartphone device with access to internet connection

Exclusion Criteria:

* Patients with cognitive impairment
* Active use of antibiotics at the time of stool collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have consented to the Mayo Clinic Biobank with gastrointestinal disease.
Sampling Method: Non-Probability Sample
Enrollment: 4001 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To Correlate Differences in Diet and Microbiome with Different GI Symptoms and Disease States | From enrollment through study completion, an average of 1 year.
  Investigators will prospectively follow the clinical course of the patients throughout the duration of the study. Patient health outcomes will be documented from their medical record while the study is actively enrolling or undergoing data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Purna Kashyap, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asnicar F, Berry SE, Valdes AM, Nguyen LH, Piccinno G, Drew DA, Leeming E, Gibson R, Le Roy C, Khatib HA, Francis L, Mazidi M, Mompeo O, Valles-Colomer M, Tett A, Beghini F, Dubois L, Bazzani D, Thomas AM, Mirzayi C, Khleborodova A, Oh S, Hine R, Bonnett C, Capdevila J, Danzanvilliers S, Giordano F, Geistlinger L, Waldron L, Davies R, Hadjigeorgiou G, Wolf J, Ordovas JM, Gardner C, Franks PW, Chan AT, Huttenhower C, Spector TD, Segata N. Microbiome connections with host metabolism and habitual diet from 1,098 deeply phenotyped individuals. Nat Med. 2021 Feb;27(2):321-332. doi: 10.1038/s41591-020-01183-8. Epub 2021 Jan 11. PMID 33432175
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Background] Thaiss CA, Itav S, Rothschild D, Meijer MT, Levy M, Moresi C, Dohnalova L, Braverman S, Rozin S, Malitsky S, Dori-Bachash M, Kuperman Y, Biton I, Gertler A, Harmelin A, Shapiro H, Halpern Z, Aharoni A, Segal E, Elinav E. Persistent microbiome alterations modulate the rate of post-dieting weight regain. Nature. 2016 Dec 22;540(7634):544-551. doi: 10.1038/nature20796. Epub 2016 Nov 24. PMID 27906159
- [Background] Sudharsan B, Peeples M, Shomali M. Hypoglycemia prediction using machine learning models for patients with type 2 diabetes. J Diabetes Sci Technol. 2015 Jan;9(1):86-90. doi: 10.1177/1932296814554260. Epub 2014 Oct 14. PMID 25316712
- [Background] Fallaize R, Macready AL, Butler LT, Ellis JA, Lovegrove JA. An insight into the public acceptance of nutrigenomic-based personalised nutrition. Nutr Res Rev. 2013 Jun;26(1):39-48. doi: 10.1017/S0954422413000024. Epub 2013 Apr 8. PMID 23561449
- [Background] Berry SE, Valdes AM, Drew DA, Asnicar F, Mazidi M, Wolf J, Capdevila J, Hadjigeorgiou G, Davies R, Al Khatib H, Bonnett C, Ganesh S, Bakker E, Hart D, Mangino M, Merino J, Linenberg I, Wyatt P, Ordovas JM, Gardner CD, Delahanty LM, Chan AT, Segata N, Franks PW, Spector TD. Human postprandial responses to food and potential for precision nutrition. Nat Med. 2020 Jun;26(6):964-973. doi: 10.1038/s41591-020-0934-0. Epub 2020 Jun 11. PMID 32528151
- [Background] Albers DJ, Levine M, Gluckman B, Ginsberg H, Hripcsak G, Mamykina L. Personalized glucose forecasting for type 2 diabetes using data assimilation. PLoS Comput Biol. 2017 Apr 27;13(4):e1005232. doi: 10.1371/journal.pcbi.1005232. eCollection 2017 Apr. PMID 28448498
- [Background] Murayama S, Numaguchi Y, Robinson AE, Richardson DE. Magnetic resonance imaging of calvarial eosinophilic granuloma. J Comput Tomogr. 1988 Oct;12(4):251-2. doi: 10.1016/0149-936x(88)90078-1. PMID 3197424
- [Background] GBD 2017 Diet Collaborators. Health effects of dietary risks in 195 countries, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 May 11;393(10184):1958-1972. doi: 10.1016/S0140-6736(19)30041-8. Epub 2019 Apr 4. PMID 30954305